CLINICAL TRIAL: NCT02780895
Title: Human OK99 Allogeneic Stem Cell Transplantation for Patients With Severe Parkinson's Disease
Brief Title: Parkinsonian Brain Repair Using Human Stem Cells
Acronym: HSCfPD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celavie Bioscences, LLC (Industry)
Collaborators: Hospital Angeles del Pedregal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OK99-2014-2017; CMN2012-027 (Other: COFEPRIS Federal Commission for the Protection against Sanitary Risk (Mexico))
Record Dates: First submitted 2016-05-12; First posted 2016-05-24 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Parkinson Disease; stereotactic surgery; human allogeneic fetal derived stem cells
MeSH Terms: conditions — Parkinson Disease | interventions — TNK1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental): stereotactic brain surgery of human stem cells (OK99)
  Interventions: Drug: Human Stem Cells

INTERVENTIONS:
Drug: Human Stem Cells — MRI-guided stereotactic intraputaminal cell implantation into PD patients was performed.
  For target locations, measurements were made using CT-scan images fused with previous MR images. Bilateral parasagittal incisions and corresponding 14 mm burr holes were made in preparation for cell suspension injections.
  To ensure complete cell suspension delivery, injections were carried out slowly for 2 min with reciprocal withdrawal of the delivery needle to avoid both damage to stem cells and brain tissue, as well as to avert reflux or bubble formation.
  After surgery, patients were kept in a conventional post-operative care unit for 1 h. The day following surgery, MR images were obtained to confirm correct placement of cell suspensions. All patients were discharged 24 h after surgery.
  Other Names: OK99

SUMMARY:
Implantation of Celavie human stem cells (OK99) is intended to address the underlying pathology of the disease by replacing damaged/destroyed cells of the brain, and/or stimulating the patient's brain to repair itself.

DETAILED DESCRIPTION:
This trial is a longitudinal, prospective, interventional, uncontrolled study designed to test, firstly, the safety and secondly, the potential efficacy of intraputaminal grafting of undifferentiated hfSC for the treatment of PD. Patients were monitored carefully for any adverse effects. All patients underwent baseline and 6- and 12-month post-surgery neurological, neuropsychological, MRI, and PET evaluations.

Procurement, isolation, expansion, and characterization of hfSC, as well as assessment of patients' immune response to hfSC grafting, were performed at Celavie Biosciences, LLC (Oxnard, CA USA). Patient selection, pre- and post-surgery neurological, neuropsychological, and MRI evaluations, as well as stereotactic surgery and post-surgery care, were performed at Hospital Angeles del Pedregal (Mexico City, Mexico). Synthesis of radiopharmaceuticals and PET imaging were carried out at the Radiopharmacy-Cyclotron Unit of the Faculty of Medicine, Universidad Nacional Autonoma de Mexico (Mexico City, Mexico). Eight patients with moderate to advanced PD were selected for this trial. One of the patients was lost to follow up due to reasons unrelated to this study. Subjects that completed follow up were 2 females and 5 males, with ages ranging between 43-74 years (mean age 56 years).

Procurement and expansion of hfSC

Human fetal brain tissue was procured via routine sterile manual aspiration methods with informed consent from the donor in accordance with NIH guidelines for use of fetal tissue as well as federal, and state laws. Tissue donor and hfSC recipients remained unknown to each other.

Maternal blood samples (sera) were tested for: HIV (Abbott Laboratories, Abbott Park IL, USA) hepatitis A, B and C (Abbott); HTLVI (Abbott); VDRL (Baxter Agglutination Slide Test and reflex FTA), and cytomegalovirus (Quest, Oxnard CA). Women with a history of genital herpes, cancer, asthma, lupus, rheumatoid arthritis, allergies, vasculitis of autoimmune origin, and drug abuse were excluded. Gestation was determined according to Carnegie stages. Fetal tissue was harvested at the sixth week of gestation after elective abortion. Fetal brain was dissected, minced and triturated to a single cell suspension. Cells were cultured in flasks incubated at 37°C under hypoxic conditions (5% O2 and 5% CO2) through 4 doublings. At the second doubling (D2) cell culture was tested for sterility (USP <71>) and at D4 culture was karyotyped and PCR tested for presence of adventitious agents: HTLV-1, HTLV-2, HIV-1 (A, B, D, F, H, N), hepatitis A, B and C, T. p. pallidum, CMV, HSV-1, HSV-2, HPV. Cells were then transferred to a closed bioreactor system (GE WAVE Bioreactor 2/10 System, Uppsala SWE), operating under the same physical and chemical conditions. The bioreactor was used to create the Master Cell Bank (MCB), which was harvested, tested, characterized and rate-control cryopreserved after a total of seven doublings (D7).

After the MCB was safety tested and characterized, a portion of the batch was thawed and used to seed the bioreactor for the Working Cell Bank (WCB) production. Cells were cultured in the bioreactor until they reached D13. They were harvested (Centritech LAB-III, Carr Centritech Separation System, Rancho Cucamonga, CA, USA), aliquoted (Fill-It; TAP Biosystems, Wilmington, DE, USA), and cryopreserved to create a WCB. The WCB was subjected to release testing for safety and characterization assays. Safety testing included sterility (USP <71>), mycoplasma (USP <63), endotoxin (USP <85>), and karyotyping (Cell Line Genetics, Madison WI, USA). Characterization included flow cytometry testing for: Oct-4 >90% (10H11.2, EMD Millipore, Billerica, MA, USA; AF488 conjugated), Sox-2 >90% (Btjce, eBioscience, San Diego CA, USA; AF488 conjugated), MHC-I <10% (A4, eBioscience; APC conjugated), MHC-II <10% (CVS20, Novus Biologicals, Littleton CO, USA; AF488 conjugated), CD105 <10% (SN6, eBioscience; PE-Cy7 conjugated), and tyrosine hydroxylase <10% (EP1532Y, Abcam, Cambridge, UK; FITC conjugated goat anti-rabbit IgG; Abcam; polyclonal). Both MCB and WCB were stored in gas phase LN2 at -196°C.

All procedures were performed under aseptic conditions in an ISO 8 clean room, utilizing ISO 5 bio-safety cabinets and laminar airflow hoods, according to validated protocols. Cells were shown to have a normal karyotype and did not produce teratomas in immunocompromised rodents (unpublished data).

Pharmacotherapy

Immunosuppression via cyclosporine A at a dose of 15 mg/kg/day was started 10 days prior to surgery and continued for one month thereafter. Patients also received Indomethacin 225mg/day, starting at 10 days prior to implantation and for six months postoperatively thereafter. Wide spectrum antibiotic (Zannat 700mg) was given preoperatively and 48 hours post-operatively. Antiparkinsonian medications were adjusted to patient's requirements.

Stereotactic surgery

MRI-guided stereotactic intraputaminal cell implantation into PD patients was performed using a Leksell Stereotactic System and Stealth Station Surgical Navigation System (Fridley, Minnesota, USA). Ropivacaine was used as a local anesthetic for frame placement. For target locations, measurements were made using CT-scan images fused with previous MR images (both in DICOM format, in axial sections 1.0 mm thick). With the patient under general anesthesia, the stereotactic frame was fixed to the operating table with a Mayfield head holder. Bilateral parasagittal incisions and corresponding 14 mm burr holes (one for each hemisphere) were made in preparation for cell suspension injections. Two different needle tracks through the same burr hole were selected for each side. Target locations were determined by height and length of putaminal nuclei. The lowest Z-coordinates of each track were located in the dorsal putamen and spaced 4mm apart in the X-direction. Each needle track received 1X106 cells in 1 cc of culture medium. To ensure complete cell suspension delivery, injections were carried out slowly for 2 min with reciprocal withdrawal of the delivery needle to avoid both damage to stem cells and brain tissue, as well as to avert reflux or bubble formation. After surgery, patients were kept in a conventional post-operative care unit for 1 h. The day following surgery, MR images were obtained to confirm correct placement of cell suspensions. All patients were discharged 24 h after surgery.

Neurological evaluations

Neurological endpoints of this study included evaluation of the number and severity of adverse events after cell grafting, and the efficacy in the improvement of motor responses, as assessed on the UPDRS part I (mentation, behavior and mood), part II (motor activities of the daily living), part III (motor performance), and part IV (complications of therapy), as well as the modified Höehn and Yahr Scale, and the modified Schwab and England Activities of the Daily Living Scale. Patients were clinically evaluated with these scales at screening (as baseline, before surgery), and then after the procedure at six and 12 months. At every visit, patients were asked to discontinue antiparkinsonian medications at least 12 hours before the UPDRS assessment (for practical purposes, "OFF" state was defined as overnight drug withdrawal) in order to be rated in their "OFF" state and then, UPDRS "ON" medication evaluations were performed 1 hour after receiving their usual dose of levodopa. Each patient received the same preoperative levodopa dose for each assessment. Adverse events, including those reported by the patients spontaneously and those observed during the evaluations were recorded. After obtaining signed informed consent from all patients that completed the study, all "OFF" and "ON" UPDRS evaluations, were videotaped.

Neuropsychological evaluations

Cognitive performance was evaluated using the following instruments: Mexican adaptations of Beck and Steer's anxiety [25] and depression [26] inventories; our brief neuropsychological (NEUROPSI)[27,28] and computerized neuropsychological test batteries, and the Mini-mental Parkinson State Examination (MMPSE)[29]. Patients reported on their quality of life as related to their daily living activities; physical and mental well-being (health status); cognition and communication, and one summary index.

Immunogenicity testing

Patient's blood was evaluated for increase in titers of hfSC specific antibodies and for increase in antibody-dependent cell-mediated cytotoxicity after implantation as compared to baseline values. Samples were drawn one month prior to cell implantation, and then one month and six months after surgery. Whole blood specimens were collected from each patient and processed as serum one and six months post-grafting using the lipophilic membrane dye PKH67 (Sigma-Aldrich) as described by the manufacturer for cell tracking in immune response and cytotoxicity assays by flow cytometry [30,31]. Cytotoxicity assay was performed with 100:1, 50:1, and 25:1 effector to target ratios.

MRI

MR images were obtained before surgery (baseline) and three times after cell implantation at 24 h, and six and 12 months post-surgery. They were acquired with a 3 Tesla magnet, MR Systems Achieva release 2.6.3.8 Philips (Best, The Netherlands).

PET molecular imaging

Patients underwent PET molecular imaging at baseline, at six months (data not presented), and at one year after hfSC implantation. Radiopharmaceuticals utilized were (+)-alpha-[11C]Dihidrotetrabenazine (DTBZ), 6-[18F]Fluoro-L-DOPA (FDOPA), and [11C]Raclopride (RAC). All patients underwent DTBZ-PET scans and one additional study with either FDOPA or RAC, at least one week apart. Patients were asked to discontinue antiparkinsonian medications at least 12h before each study. Scans were acquired on a Siemens Biograph 64 PET/CT. Thirty-minute brain emission scans were acquired 20 minutes post-injection of DTBZ or RAC, while 15 min scans were acquired for FDOPA 75 min post-injection. All patients studied with FDOPA were pre-medicated with 150 mg of carbidopa to prevent peripheral decarboxylation. Images were reconstructed using an OSEM-2D algorithm and analyzed with the software Statistical Parametric Mapping (SPM v.12). Each individual PET brain image was normalized on an anatomical MRI atlas to be evaluated within a standard space. Following normalization, FSL structural atlases were used for definition of the regions of interest. To facilitate the quantitative analysis, specific uptake ratios (SUR) in the caudate and putamen were calculated by subtracting the background signal of a reference region with nonspecific uptake from striatal activity and dividing by reference region activity [(target uptake - reference uptake)/reference uptake], using occipital cortex (DTBZ and FDOPA) and cerebellum (RAC), as reference regions.

Statistical analysis

Comparisons between baseline and 12-month follow-up measurements for anxiety, depression, NEUROPSI, MMPSE examinations, right and left finger tapping in "ON" and "OFF" medication states were performed using the Wilcoxon test. All other end measures were reported as individual results for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD with tremor, rigidity or hypokinesia as major symptoms.
* A two to twenty-five-year history of PD with significant medical management or difficulty in medical management.
* A definite response to levodopa compounds with inadequately relieved of symptoms, or severe secondary effects of the drug.
* Good general health.
* A strong will or desire to have the procedure after being fully informed of its experimental nature.

Exclusion Criteria:

* History of repeated strokes with stepwise progression of parkinsonian features
* History of repeated head injury
* History of definite encephalitis
* Oculogyric crises (unless drug-induced)
* Neuroleptic treatment at onset of symptoms
* Supranuclear gaze palsy
* Cerebellar signs
* Babinski sign
* Presence of cerebral tumor or communicating hydrocephalus on CT scan
* Sustained remission or negative response to an adequate dose of levodopa
* Patients with parkinsonism other than Idiopathic PD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety as Measured by the Number and Severity of Adverse Events | three years

SECONDARY OUTCOMES:
FDOPA (L-3,4-dihydroxy-6-(18)F-fluorophenylalanine) uptake | three years
  Positron Emission Tomography
Raclopride uptake | three years
  Positron Emission Tomography
DTBZ ([18F]9-fluoropropyl-(+)-dihydrotetrabenazine) uptake | three years
  Positron Emission Tomography
Barona Demographic Equation | three years
  Premorbid Estimates
North American Adult Reading Test (NAART) | three years
  Premorbid Estimates
Wechsler Test of Adult Reading (WTAR) | three years
  Premorbid Estimates
Wide Range AchievementTest (WRAT) | three years
  Premorbid Estimates
Mattis Dementia Rating Scale (DRS) | three years
  Neuropsychological Screening
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | three years
  Neuropsychological Screening
Intelligence Kaufman Brief Intelligence Test (KBIT) | three years
  Neuropsychological Screening
Raven's Progressive Matrices | three years
  Neuropsychological Screening
Wechsler Abbreviated Scale of Intelligence (WASI) | three years
  Neuropsychological Screening
Wechsler Adult Intelligence Scale (WAIS) | three years
  Neuropsychological Screening
Auditory Consonant Trigrams (ACT) | three years
  Attention and Working Memory
Brief Test of Attention (BTA) | three years
  Attention and Working Memory
Continuous Performance Tests (CPT) | three years
  Attention and Working Memory
Digit and Visual Spans | three years
  Attention and Working Memory
Paced Auditory Serial Addition Test (PASAT) | three years
  Attention and Working Memory
Stroop Test | three years
  Attention and Working Memory
Cognitive Estimation Test (CET) | three years
  Executive Function
Delis-Kaplan Executive Function Scale (DKEFS) | three years
  Executive Function
Halstead Category Test | three years
  Executive Function
Trailmaking Test (TMT) | three years
  Executive Function
Wisconsin Card Sorting Test (WCST) | three years
  Executive Function
Benton Visual Retention Test (BVRT-R) | three years
California Verbal Learning Test (CVLT) | three years
  Memory
Rey Auditory Verbal Learning Test (RAVLT) | three years
  Memory
Rey Complex Figure Test (RCFT) | three years
  Memory
Wechsler Memory Scale (WMS) | three years
  Memory
Boston Naming Test (BNT) | three years
  Language
Controlled Oral Word Association Test (COWAT) | three years
  Language
Sentence Repetition | three years
  Language
Token Test | three years
  Language
Complex Ideational Material | three years
  Language
Benton Facial Recognition Test | three years
  Visuoperception
Benton Judgment of Line Orientation (JLO) | three years
  Visuoperception
Hooper Visual Organization Test (VOT) | three years
  Visuoperception
Finger Tapping | three years
  Motor and Sensory Perception
Grooved Pegboard | three years
  Motor and Sensory Perception
Hand Dynamometer | three years
  Motor and Sensory Perception
Sensory-Perceptual Examination | three years
  Motor and Sensory Perception
Beck Anxiety Inventory (BAI) | three years
  Mood State and Personality
Beck Depression Inventory (BDI) | three years
  Mood State and Personality
Hamilton Depression Scale (HDS) | three years
  Mood State and Personality
Minnesota Multiphasic Personality Inventory (MMPI) | three years
  Mood State and Personality
Proﬁle of Mood States (POMS) | three years
  Mood State and Personality
State-Trait Anxiety Inventory (STAI) | three years
  Mood State and Personality
Parkinson's Disease Questionnaire (PDQ) | three years
  Quality of Life, Coping, and Stressors
Coping Responses Inventory (CRI) | three years
  Quality of Life, Coping, and Stressors
Ways of Coping Questionnaire | three years
  Quality of Life, Coping, and Stressors
Life Stressors and Social Resources Inventory (LISRES) | three years
  Quality of Life, Coping, and Stressors
Efficacy as measured by the Unified Parkinson Disease Rating Scale (UPDRS) | three years

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Kopyov, MD, PhD, Study Director — Celavie Bioscences, LLC; Ignacio Madrazo, MD, PhD, Principal Investigator — Hospital Angeles del Pedregal
Locations (1):
- Hospital Angeles del Pedregal, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes